CLINICAL TRIAL: NCT02617758
Title: An Open-Label, Randomized, Single Application, Two-Period Crossover, Pivotal Bioequivalence Study to Evaluate the Bioequivalence of Fentanyl Transdermal System (JNJ-35685-AAA-G021) Compared With DURAGESIC Fentanyl Transdermal Patch in Healthy Subjects
Brief Title: Bioequivalence Study of Fentanyl Transdermal System (JNJ-35685-AAA-G021) Compared With DURAGESIC Fentanyl Transdermal Patch in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CR108059; FENPAI1023 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2015-11-17; First posted 2015-12-01 (Estimated); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Healthy
Keywords: Healthy; Bioequivalence Study; JNJ-35685-AAA-G021; DURAGESIC
MeSH Terms: interventions — Fentanyl

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes

ARMS (2):
- Treatment AB (Experimental): Participants will receive Treatment A (single application of DURAGESIC fentanyl transdermal system 100 microgram per hour (µg/h) dose) as Reference in Period 1; followed by Treatment B (single application of Fentanyl transdermal system [JNJ-35685-AAA-G021] 100 µg/h dose) as test in Period 2. A washout period of at least 8 days and no more than 14 days will be maintained between each treatment period.
  Interventions: Drug: Fentanyl
- Treatment BA (Experimental): Participants will receive Treatment B [single application of Fentanyl transdermal system (JNJ-35685-AAA-G021) 100 microgram per hour (µg/h) dose] as test in Period 1; followed by Treatment A (single application of DURAGESIC fentanyl transdermal system 100 µg/h dose) as Reference in Period 2. A washout period of at least 8 days and no more than 14 days will be maintained between each treatment period.
  Interventions: Drug: Fentanyl

INTERVENTIONS:
Drug: Fentanyl — Participants will receive single application of DURAGESIC fentanyl transdermal system 100 µg/h dose in one of the treatment periods.
  Other Names: DURAGESIC
Drug: Fentanyl — Participants will receive single application of Fentanyl transdermal system (JNJ-35685-AAA-G021) 100 microgram per hour (µg/h) dose in one of the treatment periods.
  Other Names: JNJ-35685-AAA-G021

SUMMARY:
The purpose of this study is to evaluate the bioequivalence of the new formulation of fentanyl transdermal system (JNJ-35685-AAA-G021) compared with DURAGESIC fentanyl in healthy participants.

DETAILED DESCRIPTION:
This is a single-center, randomized (study medication assigned to participants by chance), open-label (all people know the identity of the intervention), single application and 2-way Crossover (the same medications provided to all participants but in different sequence) pivotal study to determine the bioequivalence of marketed reference formulation DURAGESIC and the test formulation Fentanyl transdermal system (JNJ-35685-AAA-G021). Approximately 56 healthy participants will participate in this study. Participants will be randomly assigned to 1 of 2 treatment sequences. The study will consist of 3 parts: Screening Phase (within 21 days before the first study drug administration of the first period), an open-label treatment Phase consisting of 2 single-application treatment periods (26 days) and End-of-Study (at the end of Period 2). The total study duration for each participant will be from 43 days to a maximum of 59 days. Participants will receive a single application 100 microgram per hour (mcg/h) dose of DURAGESIC fentanyl transdermal system as Treatment A (Reference) and 100 mcg/h Fentanyl transdermal system (JNJ-35685-AAA-G021) as Treatment B (Test). Bioequivalence will be primarily evaluated by pharmacokinetic parameters. Participants' safety will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Participant must be healthy on the basis of physical examination, medical history, vital signs, and 12-lead electrocardiogram (ECG) performed at Screening. This determination must be recorded in the participant's source documents and initialed by the investigator
* Not of childbearing potential: postmenopausal [greater than (>) 45 years of age with amenorrhea for at least 12 months; permanently sterilized (example, bilateral tubal occlusion [which includes tubal ligation procedures as consistent with local regulations], hysterectomy, bilateral salpingectomy, bilateral oophorectomy); or otherwise be incapable of pregnancy
* Of childbearing potential and practicing a reliable method of birth control, throughout the study and for 1 week after the study is completed. The method must be consistent with local regulations regarding the use of birth control methods for participants participating in clinical studies: example, established use of oral, injected or implanted hormonal methods of contraception; placement of an intrauterine device (IUD) or intrauterine system (IUS); double-barrier methods: condom with spermicidal foam/gel/film/cream/suppository or occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/suppository; male partner sterilization (the vasectomized partner should be the sole partner for that participant); true abstinence (when this is in line with the preferred and usual lifestyle of the participant)
* A woman of childbearing potential must have a negative serum (beta-human chorionic gonadotropin [beta-hCG]) test at Screening and urine pregnancy test at Day -1 of the first treatment period
* A man who is sexually active with a woman of childbearing potential and has not had a vasectomy must agree to use a barrier method of birth control example, either condom with spermicidal foam/gel/film/cream/suppository or partner with occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/suppository, and all men must also not donate sperm during the study and for 3 months after completion of the study
* Participant must be willing and able to adhere to the prohibitions and restrictions as specified in the protocol

Exclusion Criteria:

* Participant has a history of or current clinically significant medical illness including but not limited to, cardiac arrhythmias or other cardiac disease; hematologic disease; coagulation disorders (including any abnormal bleeding or blood dyscrasias); lipid abnormalities; significant pulmonary disease, including bronchospastic respiratory disease; diabetes mellitus; hepatic or renal insufficiency [(creatinine clearance below 60 milliliter per minute (mL/min)]; thyroid disease; neurologic or psychiatric disease; infection; or any other illness that the investigator considers should exclude the participant or that could interfere with the interpretation of the study results
* Clinically significant abnormal values for hematology, clinical chemistry, or urinalysis at Screening as deemed appropriate by the investigator
* Clinically significant abnormal physical examination, vital signs or 12 lead ECG at Screening as deemed appropriate by the investigator
* Use of medications or treatments that would significantly influence or exaggerate patch adhesion or that would alter inflammatory or immune response to the study product [example, antihistamines, systemic or topical corticosteroids, cyclosporine, tacrolimus, cytotoxic drugs, immune globulin, Bacillus Calmette-Guerin (BCG), monoclonal antibodies, radiation therapy]. Throughout the study, prescription or nonprescription medication (including vitamins and herbal supplements) other than the study drugs [Fentanyl Transdermal Therapeutic System (TTS), Naloxone and Naltrexone] are prohibited, except for acetaminophen and hormonal contraceptives by women participants. The use of acetaminophen is allowed until 3 days before each study drug administration. Throughout the study, a maximum of 3 doses per day of 325 milligram (mg) acetaminophen, and no more than 3 gram (g) during the time of confinement of each dosing period will be allowed for the treatment of headache or other pain
* History of drug or alcohol abuse according to Diagnostic and Statistical Manual of Mental Disorders (4th edition) criteria within 5 years before Screening or positive test result(s) for alcohol and/or drugs of abuse (such as barbiturates, cannabinoids, alcohol, opiates, cocaine, amphetamines, benzodiazepines, hallucinogens (phencyclidine, psilocybin, and d-lysergic acid diethylamide [LSD]), or barbiturates at Screening

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2015-11 (Actual); Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Maximum Plasma Concentration (Cmax) of Fentanyl | Pre-dose; 0.5, 1, 2, 3, 5, 8, 12, 18, 24, 30, 36, 42, 48, 54, 60, 66, 72, 73, 74, 78, 84, 94, 108 and 120 hours post-dose on Day 1 of each period
  The Cmax is the maximum observed plasma concentration of Fentanyl.
Time to Reach the Maximum Plasma Concentration (Tmax) of Fentanyl | Pre-dose; 0.5, 1, 2, 3, 5, 8, 12, 18, 24, 30, 36, 42, 48, 54, 60, 66, 72, 73, 74, 78, 84, 94, 108 and 120 hours post-dose on Day 1 of each period
  The Tmax is the time to reach the maximum observed plasma concentration of Fentanyl.
Area Under the Plasma Concentration-Time Curve From 0 to Last Quantifiable Concentration (AUC[0-last]) Post Dose of Fentanyl | Pre-dose; 0.5, 1, 2, 3, 5, 8, 12, 18, 24, 30, 36, 42, 48, 54, 60, 66, 72, 73, 74, 78, 84, 94, 108 and 120 hours post-dose on Day 1 of each period
  The AUC(0-last) is the area under the plasma concentration-time curve from 0 to time of the last quantifiable concentration.
Area Under the Plasma Concentration-Time Curve From 0 to Infinite Time (AUC[0-infinity]) Post Dose of Fentanyl | Pre-dose; 0.5, 1, 2, 3, 5, 8, 12, 18, 24, 30, 36, 42, 48, 54, 60, 66, 72, 73, 74, 78, 84, 94, 108 and 120 hours post-dose on Day 1 of each period
  The AUC (0-infinity) is the area under the plasma Fentanyl concentration-time curve from time 0 to infinite time, calculated as the sum of AUC (0-last) and C(last)/lambda(z), in which AUC(0-last) is area under the plasma Fentanyl concentration-time curve from time zero to time of the last quantifiable concentration, C(last) is the last observed quantifiable concentration and lambda(z) is elimination rate constant.
Terminal Half-life (t[1/2]) of Fentanyl | Pre-dose; 0.5, 1, 2, 3, 5, 8, 12, 18, 24, 30, 36, 42, 48, 54, 60, 66, 72, 73, 74, 78, 84, 94, 108 and 120 hours post-dose on Day 1 of each period
  Elimination half-life associated with the terminal slope Lambda (z) of the semi logarithmic drug concentration-time curve, calculated as 0.693/Lambda (z).

SECONDARY OUTCOMES:
Skin Adherence Score of Fentanyl Transdermal System | Up to 72 hours post-dose on Day 1 of each period
  The Food and Drug Administration (FDA) scoring system will be the basis to evaluate adhesion performance of the transdermal system. The scoring system has scale from 0-4. Where, 0 = system adhered to greater than or equal to (>=) 90 percent (%) adhered of the area, essentially no lift off the skin; 1 = system >=75% to less than (<) 90% adhered, some edges only lifting off the skin; 2 = system >=50% to <75% adhered, less than half of the patch lifting off the skin; 3 = system greater than (>) 0% to <50% adhered, more than half of the patch lifting off the skin but not falling off; 4 = system 0% adhered to skin, patch completely off the skin.
Number of Participants with Adverse Events (AEs) and Serious AEs | Screening up to End-of-Study (Approximately Day 59)
  An adverse event (AE) is any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. A serious adverse event (SAE) is an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (1):
- Cypress, California, United States